CLINICAL TRIAL: NCT06949215
Title: 68Ga-NYM096 PET/ CT for the Detection of Clear Cell Renal Cell Carcinoma in Presurgical Patients With Complex Cystic Renal Leision
Brief Title: 68Ga-NYM096 PET/ CT for the Detection of ccRCC in Presurgical Patients With Complex Cystic Renal Leision
Acronym: NYCRCCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYCRCCL
Record Dates: First submitted 2025-02-23; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: ccRCC; Complex Renal Cyst
Keywords: PET/CT; complex renal cyst; 68Ga-NYM096

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-NYM096 PET/CT (Experimental): Each patient will receive one dose of 68Ga-NYM096 by intravenous route. Dedicated whole-body PET/CT imaging will be performed.
  Interventions: Diagnostic Test: 68Ga-NYM096 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-NYM096 PET/CT — Participants will be administered a single, intravenous bolus of 68Ga-NYM096 The recommended administered activity of 68Ga-NYM096 is 1.8-2.2 MBq per kilogram bodyweight, subject to variation that may be required owing to variable elution efficiencies obtained during the lifetime of the 68Ga / 68Ga generator.
  The CT and PET imaging session will begin approximately 45 to 75 minutes after 68Ga-NYM096 administration.

SUMMARY:
This is a prospective, single-center, single-arm, diagnostic phase 2 study aimed at evaluating the sensitivity and specificity of 68Ga-NYM096 PET/CT in detecting clear cell renal cell carcinoma (ccRCC) in patients with complex renal cysts who are scheduled for surgical resection. The study will use histopathological diagnosis as the reference standard to assess the diagnostic accuracy of 68Ga-NYM096 PET/CT in identifying ccRCC within operable complex renal cystic lesion. The findings will provide critical insights into the performance of 68Ga-NYM096 PET/CT as a non-invasive imaging tool for the preoperative detection of ccRCC in this patient population.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, diagnostic phase 2 study designed to evaluate the efficacy of 68Ga-NYM096 PET/CT in detecting clear cell renal carcinoma (ccRCC) in patients with complex renal cysts who are scheduled for surgical resection. Each patient will receive a single intravenous dose of 68Ga-NYM096, followed by dedicated whole-body PET/CT imaging. Prior to tumor resection, contrast-enhanced CT imaging of the abdomen will be conducted, and if clinically indicated or as part of the local standard of care, imaging of the chest will also be performed. Both imaging modalities (68Ga-NYM096 PET/CT and diagnostic CT) will be completed before kidney resection.

The PET/CT images will be independently interpreted by two blinded readers, while the diagnostic CT images will be evaluated by one blinded reader. The interpretations from both imaging modalities will be compared with histopathologic findings to estimate sensitivity, specificity, and predictive values (primary and secondary objectives). Additionally, the study will explore the performance of 68Ga-NYM096 PET/CT in detecting metastases compared to diagnostic CT. This study aims to provide insights into the diagnostic accuracy of 68Ga-NYM096 PET/CT for identifying ccRCC in patients with complex renal cysts.

The pathologist will identify representative tumor tissue for the determination of histology, grading, and CAIX expression.

39 patients will be recruited in Peking Union Medical College Hospital. This study will be conducted according to local regulations and laws, the ethical principles that have their origin in the Declaration of Helsinki, and the principles of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y
2. Presence of complex renal cyst (Bosniak category II or higher)
3. Scheduled for surgical resection of renal mass (partial or total nephrectomy, open, laparoscopic, or robot-assisted technique)
4. Expected survival of at least 3 months
5. ECOG ≤ 2
6. Written informed consent provided for participation in the trial
7. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. On VEGF TKI treatment less than 1 week before 68Ga-NYM096 PET/CT. TKI is known to affect girentuximab binding in patients with ccRCC and is expected to have the same effect on 68Ga-NYM096. If patients were on VEGF TKI treatment, such as sunitinib, sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NYM096 PET/CT is required.
2. Intercurrent medical condition that renders the patient ineligible for surgery.
3. Pregnancy or breastfeeding.
4. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Binary reading of renal lesions identified on 68Ga-NYM096 PET/CT | From study completion to 1 month after completion
  Define lesion as PET positive or PET negative lesion. The kidney lesion is designated as positive if the SUVmax of kidney lesions is higher than that of liver (reference).
Histological classification of operated renal lesions | From study completion to 1 month after completion
  The histological classification of operated renal lesions will be determined according to WHO classification of tumors, Feb 2004.

SECONDARY OUTCOMES:
SUVmax of renal lesions identified on 68Ga-NYM096 PET/CT | From study completion to 1 month after completion
  For kidney lesions, the tracer uptake is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimensional region of interest (ROI) over the lesion using a threshold of 40% SUVmax. The ROI should be drawn with caution not to include any adjacent normal kidney parenchyma.
Intensity of CAIX staining of operated renal lesions | From study completion to 1 month after completion
  The intensity of CAIX staining of operated renal lesions will be based on a 4-point scale from 0-3 according to the method of Bui et al, 2003
SUVmax of liver uptake on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  The liver uptake (SUVmax (liver)) is used as the references to define PET positive lesions. It is measured by placing a 3-cm region of interest in right lobe at the level of porta hepatis. Focal lesion should be avoided if present.
Tumor grade of operated renal lesions | From study completion to 1 month after completion
  The tumor grade of operated renal lesions will be determined according to Fuhrmann grading system
Extent of CAIX staining of operated renal lesions | From study completion to 1 month after completion
  The extent of CAIX staining of operated renal lesions will be determined by the percentage of the target tissue sample that have positive CAIX expression according to the method of Bui et al, 2003
Binary reading of renal lesions identified on diagnostic CT | From study completion to 1 month after completion
  A tumor will be described as clear cell renal carcinoma on a triphasic CT if one of the following two parameters is applicable:
  Significant (>85 HU) enhancement in the cortico-medullary phase Significant (>45 HU) enhancement in the parenchyma / excretory phase
Size of renal lesions identified on diagnostic CT | From study completion to 1 month after completion
  The longest diameter of the tumor will be measured on diagnostic CT
Bosniak category of lesion on diagnostic CT | From study completion to 1 month after completion
  The Bosniak category of lesions on diagnostic CT will be determined by radiologist.
Number of metastatic lesions identified on 68Ga-NYM096 PET/CT | From study completion to 1 month after completion
  For metastasis evaluation, any focal accumulation of 68Ga-NYM096 outside the kidneys that cannot be explained by physiologic uptake is interpreted as focal lesion. The SUVmax and tumor-to-background should be evaluated. Surrounding tissue is the preferred background tissue. Should not available, the blood pool should be designated as background tissue. Any focal lesion identified on 68Ga-NYM096 PET will be considered to be positive for metastasis if SUVmax (lesion) is no less than SUVmax (liver) or tumor-to-background ratio is higher than 1.
Location of metastatic lesions identified on 68Ga-NYM096 PET/CT | From study completion to 1 month after completion
  For metastasis evaluation, any focal accumulation of 68Ga-NYM096 outside the kidneys that cannot be explained by physiologic uptake is interpreted as focal lesion. The SUVmax and tumor-to-background should be evaluated. Surrounding tissue is the preferred background tissue. Should not available, the blood pool should be designated as background tissue. Any focal lesion identified on 68Ga-NYM096 PET will be considered to be positive for metastasis if SUVmax (lesion) is no less than SUVmax (liver) or tumor-to-background ratio is higher than 1.
Size of metastatic lesions identified on 68Ga-NYM096 PET/CT | From study completion to 1 month after completion
  For metastasis evaluation, any focal accumulation of 68Ga-NYM096 outside the kidneys that cannot be explained by physiologic uptake is interpreted as focal lesion. The SUVmax and tumor-to-background should be evaluated. Surrounding tissue is the preferred background tissue. Should not available, the blood pool should be designated as background tissue. Any focal lesion identified on 68Ga-NYM096 PET will be considered to be positive for metastasis if SUVmax (lesion) is no less than SUVmax (liver) or tumor-to-background ratio is higher than 1.
Number of metastatic lesions identified on diagnostic CT | From study completion to 1 month after completion
  The number of metastatic lesions on diagnostic CT will be determined by radiologist according to the typical location, enhancement pattern of the lesions.
Location of metastatic lesions on diagnostic CT | From study completion to 1 month after completion
  The location of metastatic lesions on diagnostic CT will be determined by radiologist according to the typical location, enhancement pattern of the lesions.
Size of metastatic lesions on diagnostic CT | From study completion to 1 month after completion
  The size of metastatic lesions on diagnostic CT will be measured by radiologist according to the typical location, enhancement pattern of the lesions.

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol
Time Frame: Within 2 years after the publication of the main results